CLINICAL TRIAL: NCT01872377
Title: Phase I Time-to-Event Continual Reassessment (TITE-CRM) Dose Escalation Trial of CyberKnife® Stereotactic Body Radiotherapy (SBRT) Boost With Concurrent Chemoradiotherapy for Patients With Unresectable Locally Advanced Pancreatic Cancer
Brief Title: Dose Escalation Study of CyberKnife® SBRT Boost for Patients With Unresectable Locally Advanced Pancreatic Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No longer recruiting patients to this study
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20120384-01H; OTT 12-04
Record Dates: First submitted 2012-10-12; First posted 2013-06-07 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Pancreatic Carcinoma Non-resectable
Keywords: pancreas; pancreatic; unresectable; CyberKnife; SBRT

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiotherapy Boost (Experimental): All participants will receive the CyberKnife® Stereotactic Body Radiotherapy(SBRT)Boost treatment however, there are 5 dose levels that could be assigned according to Time-to-Event Continual Reassessment Method (TITE-CRM). Participants will be assigned to either receiving 6, 7, 8, 9 or 10 Gy X 3Fr.
  Interventions: Radiation: CyberKnife® Stereotactic Body Radiotherapy(SBRT)Boost

INTERVENTIONS:
Radiation: CyberKnife® Stereotactic Body Radiotherapy(SBRT)Boost — Stereotactic body radiotherapy (SBRT) is a minimally invasive treatment technique that allows for ultra-high doses of radiation to be delivered to small areas with precision. In this study all participants will receive one of 5 dose levels that will be assigned according to Time-to-Event Continual Reassessment Method (TITE-CRM). Three fractions of various dose levels would be delivered over 5 to 10 days (typically Monday, Wednesday and Friday) with at least 36 hours between two sessions. In case of technical or medical problem, the authorized total treatment time is 12 days.

SUMMARY:
Currently the standard treatment for locally advanced, unresectable pancreatic cancer consists either of chemotherapy by itself or a combination of chemotherapy plus radiation therapy or no treatment at all. Unfortunately, no treatment thus far has been able to provide patients with a consistent chance for a cure although there are rare patients who will live for many years after treatment. For most patients the chemotherapy or chemotherapy plus radiation will maintain or improve quality of life by keeping the cancer under control for a period of time.

Approximately 25-30% of patients with early pancreatic cancer who are able to have the cancer completely removed surgically will live beyond 5 years and will be considered cured. This tells us that aggressive treatment directed at the tumour in the pancreas can lead to cure. For the majority of patients who can not have an operation, giving more radiation as part of the treatment may be a strategy that results in better control of the tumour in the pancreas which may or may not result in patients living longer.

The purpose of this study is to test the safety of adding a higher dose (a "boost" dose) of radiation using a radiation unit called CyberKnife when combined with standard chemotherapy and radiation for patients with locally advanced, unresectable pancreatic cancer.

Participants on this study will receive a 'boost' dose of radiation which consists of 3 treatments over 1 week. The participants will then receive the standard of care treatment of chemotherapy and standard radiation therapy over a 5 week period, which will be followed by the conventional 20 weeks of chemotherapy alone. The participants will then be followed for progression of disease and toxicity related to the boost treatment for up to 5 years.

DETAILED DESCRIPTION:
Stereotactic body radiotherapy (SBRT) is a minimally invasive treatment technique that allows for ultra-high doses of radiation to be delivered to small areas with precision not previously possible using older equipment. The CyberKnife® Robotic Radiosurgery System (Accuray, Sunnyvale California, USA) is a radiation unit specifically designed to focus beams of radiation accurately anywhere in the body. It is able to track, detect and correct for any tumor movement during treatment by using a sophisticated image guidance system.

ELIGIBILITY:
Inclusion Criteria:

* Histological or Pathologically confirmed pancreatic adenocarcinoma
* T1 - T4 or N0-N1 pancreatic adenocarcinoma
* ECOG performance status ≤ 2
* Male and female, aged ≥ 19- 80 years
* Signed study-specific informed consent
* General condition considered feasible for radiotherapy
* INR ≤1.5 within 7 days prior to fiducial placement

Exclusion Criteria:

* Diagnosis of distant metastatic disease
* Primary tumor > 5 cm in maximum diameter on any imaging modality
* >3 involved lymph nodes as per staging CT and/or PET-CT
* Clear indication of involvement of duodenal wall on imaging or at time of endoscopy
* Evidence of peritoneal carcinomatosis, portal vein occlusion, ascites or involvement of non-regional lymph nodes
* Histology clearly other than adenocarcinoma
* Disease cannot be radiographically assessed due to patient related contraindications or due to lack of visible tumor on pre-treatment imaging
* More than 1 prior chemotherapy regimen for pancreatic cancer or treatment for >6 months
* Prior radiotherapy exposure that would overlap the anticipated study treatment fields
* Treatment with any other investigational agent, within 30 days prior to entering this study
* Prior chemotherapy for pancreatic cancer is permitted, although there should be 30 days between last dose and start of treatment on protocol
* Past or current history of other malignancies (except non-melanoma skin cancer or carcinoma in-situ of the cervix) unless in complete remission for a minimum of 2 years from treatment start
* Life expectancy < 12 months
* Inability or unwillingness to comply with the protocol
* Any medical condition which, in the opinion of the treating radiation oncologist, would make a radical course of radiotherapy to the upper abdomen unsafe
* Pregnancy or lactation
* Positive serum pregnancy test within 7 days of starting study treatment in pre-menopausal women and women < 2 years after the onset of menopause.
* Female participants that are of childbearing potential unwilling or unable to use effective means of contraception while receiving the study interventions and 30 days after receiving the last dose of study interventions
* Male participants ,unwilling or unable, or whose female partner is unwilling or unable, to use effective means of contraception while the participant is receiving the study interventions and 30 days after receiving the last dose of study interventions

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-07; Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
Toxicity defined as grade 3 or 4 gastro-intestinal or other non-haematological toxicity | up to 3 years
  Toxicity defined as grade 3 or 4 gastro-intestinal or other non-haematological toxicity felt to be related to radiotherapy to the upper abdomen, graded as per CTCAE 4.0 and occuring between 3 and 9 months post CyberKnife radiotherapy

SECONDARY OUTCOMES:
CT scans will measure tumour response | up to 7 years
  Participant recurrence free survival (RFS), progression free survival (PFS), time to recurrence (TTR), and overall survival (OS) will be measured using CT scans at 3 month intervals during the first 9 months post CyberKnife radiotherapy and then 6 month intervals during the remainder of follow up phase.
CyberKnife radiation dose measured in Gy delivered to the tumour and surrounding organs vs. the frequency of grade 3-4 toxicity defined by CTCAE v4.0 | up to 7 years
  To establish radiation dose-volume relationships for various organs and toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Pantarotto, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital Cancer Centre, Ottawa, Ontario, Canada